CLINICAL TRIAL: NCT04148391
Title: A Study to Evaluate NYX-458 in Subjects With Mild Cognitive Impairment or Mild Dementia Associated With Parkinson's Disease or Prodromal or Manifest Lewy Body Dementia
Brief Title: NYX-458 in Subjects With Mild Cognitive Impairment or Mild Dementia Due to Parkinson's Disease or Lewy Body Dementia (Cognition, Memory, Attention, Thinking)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aptinyx (Industry)
Collaborators: CogState Ltd. (Industry); Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NYX-458-2006
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Mild Cognitive Impairment; Mild Dementia; Parkinson Disease; Lewy Body Disease
MeSH Terms: conditions — Cognitive Dysfunction; Parkinson Disease; Lewy Body Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Matching placebo Capsules
  Interventions: Drug: Placebo Oral Capsule
- NYX-458 30 mg (Experimental): Single oral dose taken daily for 12 weeks.
  Interventions: Drug: NYX-458

INTERVENTIONS:
Drug: Placebo Oral Capsule — Matching placebo capsules.
  Arms: Placebo
Drug: NYX-458 — NYX-458 is a small molecule that modulates the N-methyl-D-aspartate receptor (NMDAR).
  Arms: NYX-458 30 mg

SUMMARY:
A Study to Evaluate NYX-458 in Subjects With Mild Cognitive Impairment or Mild Dementia Associated With Parkinson's Disease or Prodromal or Manifest Lewy Body Dementia

DETAILED DESCRIPTION:
The study will be a 16 to 18-week study, including a 2 to 4-week screening period, followed by a 12-week double-blind, randomized, placebo-controlled treatment Period, and a 2-week follow-up period. Subjects eligible for the study will be randomized to receive either NYX-458 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* Diagnosis of Parkinson's disease and mild cognitive impairment or mild dementia OR diagnosis of mild cognitive impairment or mild dementia with Lewy bodies
* Presence of subjective cognitive complaints by the patient
* Verifiable impairment, as defined a CGI-S (Clinical Global Impression-Severity) score of at least 3 (mildly ill).
* Score on the MoCA (Montreal Cognitive Assessment) between 15 and 25, inclusive.
* Stable anti-parkinsonian regimen (if applicable)
* Has a study partner who can accompany the subject at specified study visits

Exclusion Criteria:

* Clinically meaningful motor complications
* Current use of medications with primarily central nervous system activities
* Other clinically significant medical histories that may interfere with completing the study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in physical examination | Subjects will be followed up to 14 days post-dose
  Physical examination
Rates of adverse events and serious adverse events | Subjects will be followed up to 14 days post-dose
  Adverse events and serious adverse events
Rates of early termination due to adverse events | Subjects will be followed up to 14 days post-dose
  Early termination due to adverse events
Change from baseline in vital signs, clinical laboratory values, and electrocardiogram results | Subjects will be followed up to 14 days post-dose
  Vital signs, clinical laboratory values, and electrocardiogram results
Change from baseline dissociative effects, psychosis, and hallucinatory symptoms as measured by the Neuropsychiatric Inventory (NPI-12) | Subjects will be followed up to 14 days post-dose
  Neuropsychiatric Inventory (NPI-12) - NPI-12 assesses 12 behavioral domains common in dementia. Higher scores indicate more severe illness.
Change from baseline in suicidal ideation and behavior as measured by the Sheehan Suicidality Tracking Scale (S-STS) | Subjects will be followed up to 14 days post-dose
  Sheehan Suicidality Tracking Scale (S-STS) is a 16-item scale that assesses the seriousness of suicidality phenomena on a likert-type scale (0 to 4) ranging from 0 = not at all to 4 = extremely
Change from baseline in motor complications as measured by the Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part 4 | Subjects will be followed up to 14 days post-dose
  Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part 4 includes 6 items assessing motor complications, higher scores indicate more serious illness.
Change in total score of the Sheehan Suicidality Tracking Scale (S-STS) | Subjects will be followed up to 14 days post-dose
  Sheehan Suicidality Tracking Scale (S-STS) is a 16-item scale that assesses the seriousness of suicidality phenomena on a likert-type scale (0 to 4) ranging from 0 = not at all to 4 = extremely

SECONDARY OUTCOMES:
Change from baseline in the One Back test | Week 12
  The One Back test is a measure of working memory
Change from baseline in the Two Back test | Week 12
  The Two Back test is a measure of working memory
Change from baseline in the Groton Maze Learning Test | Week 12
  The Groton Maze Learning test is a measure of problem solving and reasoning
Change from baseline in the Identification Test | Week 12
  The Identification test is a measure of visual attention
Change from baseline in the International Shopping List Test | Week 12
  The International Shopping List test is a measure of verbal learning
Change from baseline on Continuous Paired Associate Learning Test | Week 12
  The Continuous Paired Associate Learning test is a measure of visual associate memory

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Aptinyx Clinical Site, Scottsdale, Arizona
  - Aptinyx Clinical Site, Fresno, California
  - Aptinyx Clinical Site, Simi Valley, California
  - Aptinyx Clinical Site, Boca Raton, Florida
  - Aptinyx Clinical Site, Bradenton, Florida
  - Aptinyx Clinical Site, Miami, Florida
  - Aptinyx Clinical Site, Miami Lakes, Florida
  - Aptinyx Clinical Site, Orlando, Florida
  - Aptinyx Clinical Site, Port Charlotte, Florida
  - Aptinyx Clinical Site, Port Orange, Florida
  - Aptinyx Clinical Site, Sunrise, Florida
  - Aptinyx Clinical Site, Decatur, Georgia
  - Aptinyx Clinical Site, Farmington Hills, Michigan
  - Aptinyx Clinical Site, Golden Valley, Minnesota
  - Aptinyx Clinical Site, Toms River, New Jersey
  - Aptinyx Clinical Site, Poughkeepsie, New York
  - Aptinyx Clinical Site, Asheville, North Carolina
  - Aptinyx Clinical Site, Dayton, Ohio
  - Aptinyx Clinical Site, Tulsa, Oklahoma
  - Aptinyx Clinical Site, Round Rock, Texas
  - Aptinyx Clinical Site, Sugar Land, Texas
  - Aptinyx Clinical Site, Bellevue, Washington
  - Aptinyx Clinical Site, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No